CLINICAL TRIAL: NCT00307047
Title: SPIRIT IV Clinical Trial: Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Subjects With de Novo Native Coronary Artery Lesions
Brief Title: SPIRIT IV Clinical Trial: Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-368
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
Keywords: Stents; Angioplasty; Total coronary occlusion; coronary restenosis; stent thrombosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XIENCE V® (Experimental)
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent
- TAXUS™ EXPRESS2™ (Active Comparator)
  Interventions: Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Other Names: XIENCE V® Everolimus Eluting Coronary Stent System
  Arms: XIENCE V®
Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Other Names: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System
  Arms: TAXUS™ EXPRESS2™

SUMMARY:
The purpose of the SPIRIT IV Clinical Trial is to continue to evaluate the safety and efficacy of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V®). The XIENCE V® arm will be compared to an active control, represented by the FDA-approved TAXUS® EXPRESS2™ Paclitaxel-Eluting Coronary Stent System (TAXUS®), commercially available from Boston Scientific.

TAXUS® EXPRESS2™ Paclitaxel Eluting Coronary Stent System is manufactured by Boston Scientific.

DETAILED DESCRIPTION:
The completion of the SPIRIT IV clinical trial at three years is justified by the consistent long-term clinical evidence supporting the safety and efficacy of the XIENCE V EECSS in complex, real-world patients across multiple geographies. As SPIRIT IV was designed as a continued access trial, completing the clinical follow-up at the three-year visit does not conflict with any FDA requirements. Abbott Vascular is committed to providing clinical outcomes through three years. The clinical evidence provided from across multiple geographies, in complex populations thus supports Abbott Vascular's proposal to complete the SPIRIT IV RCT at the three-year clinical follow-up.

The SPIRIT IV Clinical Trial is a randomized, active-controlled, single-blinded, multicenter clinical trial in the US that will enroll approximately 3,690 subjects (2:1 randomization XIENCE V®: TAXUS®). The trial allows the treatment of up to three de novo native coronary artery lesions, maximum of two lesion per epicardial vessel, with reference vessel diameters (RVD) ≥ 2.5 mm to ≤ 4.25 mm and lesion lengths ≤ 28 mm. (NOTE: RVD ≥ 2.5 mm to ≤ 3.75 mm until 4.0 mm TAXUS® is commercially available). All subjects will be screened per the protocol inclusion and exclusion criteria and enrolled subjects will have clinical follow-up at 30, 180, and 270 days and 1, 2, and 3 years.

ELIGIBILITY:
General Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving XIENCE V® and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure
* Subject must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia)
* Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
* Subject must agree to undergo all protocol-required follow-up procedures
* Subject must agree not to participate in any other clinical study for a period of one year following the index procedure

Angiographic Inclusion Criteria:

* Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥2.5 mm to ≤4.25 mm and treatment of up to a three de novo target lesions, maximum of two de novo target lesions per epicardical vessel. (NOTE: RVD ≥2.5 mm to ≤3.75 mm until 4.0 mm TAXUS® is commercially available)
* Target lesion(s) must measure ≤28 mm in length by visual estimation(≥3 mm of non-diseased tissue on either side of the target lesion should be covered by the study stent)
* If more than one target lesion will be treated, the RVD and lesion length of each must meet the above criteria
* If more than one target lesion will be treated, the RVD and lesion length of each must meet the above criteria
* The target lesion(s) must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1
* Non-study, percutaneous intervention for lesions in a target vessel (including side branches) is allowed if done ≥ 9 months prior to the index procedure
* Non-study percutaneous intervention for lesions in a non-target vessel involving:
* Successful and uncomplicated (visually estimated diameter stenosis < 50%, TIMI Grade 3 flow, no ECG changes, prolonged chest pain, or angiographic complications) bare-metal stent, balloon dilatation, cutting balloon, atherectomy, thrombectomy, and laser treatments are allowed if done ≥ 24 hours prior to the index procedure or during (before randomization) the index procedure. For interventions done within 24 to 48 hours prior to the index procedure, CK and CK-MB must be assessed to be < 2 times the upper limit of normal at the time of the index procedure. NOTE: Procedures within the 24 hour period preceding the index procedure are not permitted
* Unsuccessful or complicated bare-metal stent, balloon dilatation, cutting balloon, atherectomy, thrombectomy, and laser treatments are allowed if done ≥ 30 days prior to the index procedure
* Drug-eluting stent treatment is allowed if done ≥ 90 days prior to the index procedure
* Non-study, percutaneous interventions for lesion(s) in a target vessel (including side branches) or non-target vessel are allowed if done ≥ 9 months after the index procedure

General Exclusion Criteria:

* Subject has had a known diagnosis of acute myocardial infarction (AMI) preceding the index procedure (CK-MB ≥ 2 times upper limit of normal) and CK and CK-MB have not returned within normal limits at the time of procedure
* The subject is currently experiencing clinical symptoms consistent with AMI
* Subject has current unstable arrhythmias
* Subject has a known left ventricular ejection fraction (LVEF) < 30%
* Subject has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Subject is receiving or scheduled to receive anticancer therapy for malignancy within 30 days prior to or after the procedure
* Subject is receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.)
* Subject is receiving or is scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
* Subject has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated
* Elective surgery that will require discontinuing either aspirin or clopidogrel is planned within the first 9 months after the procedure
* Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
* Subject has known renal insufficiency (e.g., serum creatinine level of > 2.5 mg/dL or subject on dialysis)
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
* Subject has had a significant GI or urinary bleed within the past six months
* Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Subject has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a life expectancy of less than one year
* Subject is already participating in another clinical study that has not yet reached its primary endpoint
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. (Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure and effective contraception must be used up to 1 year following the index procedure)
* Angiographic Exclusion Criteria
* The target lesion(s) meets any of the following criteria:
* Left main coronary artery location including left main ostial location (NOTE: RCA-aorto-ostial lesions are not excluded)
* Located within 2 mm of the origin of the LAD or LCX
* Located within an arterial or saphenous vein graft or distal to a diseased (vessel irregularity per angiogram and any visually estimated diameter stenosis > 20%) arterial or saphenous vein graft
* Involves a bifurcation in which the side branch is ≥ 2 mm in diameter AND the ostium of the side branch is > 50% stenosed by visual estimation
* Involves a side branch requiring pre-dilatation
* Total occlusion (TIMI flow 0) prior to wire crossing
* Excessive tortuosity proximal to or within the lesion
* Extreme angulation (≥ 90º) proximal to or within the lesion
* Heavy calcification
* Restenotic from previous intervention
* Subject has received brachytherapy in any epicardial vessel (including side branches)
* The target vessel contains thrombus
* Another clinically significant lesion in the target vessel is present that requires or has a high probability of requiring PCI during the index procedure
* Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 9 months after the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3687 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, Principal Investigator — Columbia University
Locations (65):
- United States (65):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Inova Fairfax Hospital, Fairfax, California
  - San Diego Cardiovascular Associates, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - Good Samaritan Hospital - LA, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Sutter Medical Center of Santa Rosa, Santa Rosa, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sacred Heart Hospital, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. Francis Hospital and Health Centers, Indianapolis, Indiana
  - The Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center P.C., Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Saint Vincent Hospital, Worcester, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Bay Regional Medical Center, Bay City, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Dartmouth Hitchock Medical Center, Lebanon, New Hampshire
  - Millard Fillmore Hospital, Buffalo, New York
  - New York Presbyterian Hospital-Cornell, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Valley Hospital, Pomona, New York
  - Stony Brook Hospital and Medical Center, Stony Brook, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Presbyterian Hospital - Charlotte, Charlotte, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sisters of Charity Providence Hospitals, Columbia, South Carolina
  - St. Francis Health System, Greenville, South Carolina
  - Vanderbilt Vniversity Medical Center, Nashville, Tennessee
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Sentara Norfolk General, Norfolk, Virginia
  - St. Luke's Medical Center - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520
- [Derived] Muramatsu T, Onuma Y, van Geuns RJ, Chevalier B, Patel TM, Seth A, Diletti R, Garcia-Garcia HM, Dorange CC, Veldhof S, Cheong WF, Ozaki Y, Whitbourn R, Bartorelli A, Stone GW, Abizaid A, Serruys PW; ABSORB Cohort B Investigators; ABSORB EXTEND Investigators; SPIRIT FIRST Investigators; SPIRIT II Investigators; SPIRIT III Investigators; SPIRIT IV Investigators. 1-year clinical outcomes of diabetic patients treated with everolimus-eluting bioresorbable vascular scaffolds: a pooled analysis of the ABSORB and the SPIRIT trials. JACC Cardiovasc Interv. 2014 May;7(5):482-93. doi: 10.1016/j.jcin.2014.01.155. Epub 2014 Apr 16. PMID 24746650
- [Derived] Pervaiz MH, Sood P, Sudhir K, Hermiller JB, Hou L, Hattori K, Su X, Cao S, Wang J, Applegate RJ, Kereiakes DJ, Yaqub M, Stone GW, Cutlip DE. Periprocedural myocardial infarction in a randomized trial of everolimus-eluting and Paclitaxel-eluting coronary stents: frequency and impact on mortality according to historic versus universal definitions. Circ Cardiovasc Interv. 2012 Apr;5(2):150-6. doi: 10.1161/CIRCINTERVENTIONS.111.965566. Epub 2012 Mar 20. PMID 22438430
- [Derived] Claessen BE, Smits PC, Kereiakes DJ, Parise H, Fahy M, Kedhi E, Serruys PW, Lansky AJ, Cristea E, Sudhir K, Sood P, Simonton CA, Stone GW. Impact of lesion length and vessel size on clinical outcomes after percutaneous coronary intervention with everolimus- versus paclitaxel-eluting stents pooled analysis from the SPIRIT (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice) Randomized Trials. JACC Cardiovasc Interv. 2011 Nov;4(11):1209-15. doi: 10.1016/j.jcin.2011.07.016. PMID 22115661
- [Derived] Planer D, Smits PC, Kereiakes DJ, Kedhi E, Fahy M, Xu K, Serruys PW, Stone GW. Comparison of everolimus- and paclitaxel-eluting stents in patients with acute and stable coronary syndromes: pooled results from the SPIRIT (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (A Trial of Everolimus-Eluting Stents and Paclitaxel-Eluting Stents for Coronary Revascularization in Daily Practice) Trials. JACC Cardiovasc Interv. 2011 Oct;4(10):1104-15. doi: 10.1016/j.jcin.2011.06.018. PMID 22017936
- [Derived] Kereiakes DJ, Sudhir K, Hermiller JB, Gordon PC, Ferguson J, Yaqub M, Sood P, Su X, Yakubov S, Lansky AJ, Stone GW. Comparison of everolimus-eluting and paclitaxel-eluting coronary stents in patients undergoing multilesion and multivessel intervention: the SPIRIT III (A Clinical Evaluation of the Investigational Device XIENCE V Everolimus Eluting Coronary Stent System [EECSS] in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) and SPIRIT IV (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) randomized trials. JACC Cardiovasc Interv. 2010 Dec;3(12):1229-39. doi: 10.1016/j.jcin.2010.09.014. PMID 21232716
- [Derived] Kereiakes DJ, Cutlip DE, Applegate RJ, Wang J, Yaqub M, Sood P, Su X, Su G, Farhat N, Rizvi A, Simonton CA, Sudhir K, Stone GW. Outcomes in diabetic and nondiabetic patients treated with everolimus- or paclitaxel-eluting stents: results from the SPIRIT IV clinical trial (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System). J Am Coll Cardiol. 2010 Dec 14;56(25):2084-9. doi: 10.1016/j.jacc.2010.10.006. PMID 21144968
- [Derived] Stone GW, Rizvi A, Newman W, Mastali K, Wang JC, Caputo R, Doostzadeh J, Cao S, Simonton CA, Sudhir K, Lansky AJ, Cutlip DE, Kereiakes DJ; SPIRIT IV Investigators. Everolimus-eluting versus paclitaxel-eluting stents in coronary artery disease. N Engl J Med. 2010 May 6;362(18):1663-74. doi: 10.1056/NEJMoa0910496. PMID 20445180
- [Derived] Nikolsky E, Lansky AJ, Sudhir K, Doostzadeh J, Cutlip DE, Piana R, Su X, White R, Simonton CA, Stone GW. SPIRIT IV trial design: a large-scale randomized comparison of everolimus-eluting stents and paclitaxel-eluting stents in patients with coronary artery disease. Am Heart J. 2009 Oct;158(4):520-526.e2. doi: 10.1016/j.ahj.2009.07.025. Epub 2009 Aug 26. PMID 19781409

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled into this trial were comprised of male and female subjects from the general interventional cardiology population. Recruitment may have, but was not limited to a hospital or an interventional cardiology clinic. The enrollment period was August 10, 2006 through July 30, 2008.
Pre-assignment Details: Patients who met inclusion/exclusion criteria were offered participation in the study, and randomized until the total trial population was reached.
Groups:
- XIENCE V®: Patients recieving the XIENCE V® stent
- TAXUS™ EXPRESS 2™: Patients receiving the TAXUS™ EXPRESS 2™ stent
Period: Overall Study
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Started | 2458 | 1229
Completed | 2389 | 1180
Not Completed | 69 | 49
Not completed — Lost to Follow-up | 35 | 24
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Physician Decision | 1 | 2
Not completed — Lost to follow-up for other reasons | 0 | 1
Not completed — All death, all MI, all Revascularization | 27 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™ | Total
Number analyzed (Participants) | 2458 | 1229 | 3687
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1373 | 677 | 2050
  >=65 years | 1085 | 552 | 1637
Age Continuous [Mean (Standard Deviation); unit: years] | 63.25 (10.52) | 63.34 (10.23) | 63.28 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 793 | 396 | 1189
  Male | 1665 | 833 | 2498
Region of Enrollment [Number; unit: participants]
  United States | 2458 | 1229 | 3687

OUTCOME MEASURES:

1. Secondary Outcome: Ischemia Driven Target Vessel Failure (TVF)
Description: Defined as the composite endpoint comprised of cardiac death (CD), myocardial infarction (MI), TLR, and TVR
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
percentage of participants | 1.9 | 3.1

2. Secondary Outcome: Ischemia Driven Target Vessel Failure (TVF)
Description: Defined as the composite endpoint comprised of cardiac death (CD), myocardial infarction (MI), TLR, and TVR
Time Frame: 180 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
percentage of participants | 3.4 | 6.2

3. Secondary Outcome: Ischemia Driven Target Vessel Failure (TVF)
Description: Defined as the composite endpoint comprised of cardiac death (CD), myocardial infarction (MI), TLR, and TVR
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
percentage of participants | 4.6 | 7.2

4. Secondary Outcome: Ischemia Driven Target Vessel Failure (TVF)
Description: Defined as the composite endpoint comprised of cardiac death (CD), myocardial infarction (MI), TLR, and TVR
Time Frame: 1 year
Population: ITT, @ 1 yr
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
percentage of participants | 5.6 | 7.9

5. Secondary Outcome: Ischemia Driven Target Vessel Failure (TVF)
Description: Defined as the composite endpoint comprised of cardiac death (CD), myocardial infarction (MI), TLR, and TVR
Time Frame: 2 years
Population: ITT, @ 2 years
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
percentage of participants | 9.6 | 11.8

6. Secondary Outcome: Ischemia Driven Target Vessel Failure (TVF)
Description: Defined as the composite endpoint comprised of cardiac death (CD), myocardial infarction (MI), TLR, and TVR
Time Frame: 3 years
Population: ITT, @ 3 years
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
percentage of participants | 13.3 | 14.5

7. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (TLR)
Description: Revascularization of a target lesion associated with any of the following:
  * positive functional ischemia study
  * ischemic symptoms and angiographic minimal lumen diameter stenosis ≥ 50% by core laboratory quantitative coronary angiography (QCA)
  * angiographic diameter stenosis ≥ 70% by core laboratory QCA without either ischemic symptoms or a positive functional study
Time Frame: 30 days
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
percentage of participants | 0.4 | 1.1

8. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (TLR)
Description: as for outcome 7
Time Frame: 180 days
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
percentage of participants | 1.1 | 3.2

9. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (TLR)
Description: as for outcome 7
Time Frame: 270 days
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
percentage of participants | 1.9 | 4.1

10. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (TLR)
Description: as for outcome 7
Time Frame: 1 year
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
percentage of participants | 2.5 [1.94 to 3.23] | 4.6 [3.49 to 5.95]

11. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (TLR)
Description: as for outcome 7
Time Frame: 2 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
percentage of participants | 4.4 | 6.9

12. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (TLR)
Description: as for outcome 7
Time Frame: 3 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
percentage of participants | 6.3 | 7.9

13. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (TVR)
Description: Revascularization of a lesion within the target vessel associated with any of the following:
  * positive functional ischemia study
  * ischemic symptoms and an angiographic minimal lumen diameter stenosis ≥ 50% by core laboratory quantitative coronary angiography (QCA)
  * angiographic diameter stenosis ≥ 70% by core laboratory QCA without either ischemic symptoms or a positive functional study
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
percentage of participants | 0.7 | 1.6

14. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (TVR)
Description: as for outcome 13
Time Frame: 180 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
percentage of participants | 1.9 | 4.3

15. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (TVR)
Description: as for outcome 13
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
percentage of participants | 3.0 | 5.3

16. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (TVR)
Description: as for outcome 13
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
percentage of participants | 3.9 | 5.9

17. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (TVR)
Description: as for outcome 13
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
percentage of participants | 7.0 | 8.9

18. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (TVR)
Description: as for outcome 13
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
percentage of participants | 10.1 | 10.6

19. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Events (MACE)
Description: Patients determined to have had a MACE event, defined as one of the following events: Cardiac death, myocardial infarction, and TLR
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
Percentage of participants | 1.6 | 2.7

20. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Events (MACE)
Description: as for outcome 19
Time Frame: 180 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
Percentage of participants | 2.6 | 5.3

21. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Events (MACE)
Description: as for outcome 19
Time Frame: 270 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
Percentage of participants | 3.5 | 6.2

22. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Events (MACE)
Description: as for outcome 19
Time Frame: 1 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
Percentage of participants | 4.2 | 6.9

23. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Events (MACE)
Description: as for outcome 19
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
Percentage of participants | 7.2 | 10.2

24. Secondary Outcome: Ischemia Driven Major Adverse Cardiac Events (MACE)
Description: as for outcome 19
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
Percentage of participants | 9.8 | 12.3

25. Secondary Outcome: Acute Success (Clinical Device)
Description: Successful delivery and deployment of the first implanted study stent (in overlapping stent setting a successful delivery and deployment of the first and second study stents) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of final residual stenosis of less than 50% of the target lesion by QCA (by visual estimation if QCA unavailable). Bailout subjects will be included as device success only if the above criteria for clinical device are met.
Time Frame: Acute: At time of index procedure
Population: clinical device success is computed per lesion
Measure: Number; unit: Percent of success
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 3058 | 1551
Percent of success | 92.0 | 90.7

26. Secondary Outcome: Acute Success (Clinical Procedure)
Description: Successful delivery and deployment of the study stent or stents at the intended target lesion and successful withdrawal of the stent delivery system with attainment of final residual stenosis of less than 50% of the target lesion by QCA (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of major adverse cardiac event (MACE) during the hospital stay with a maximum of first seven days following the index procedure. In multiple lesion setting all lesions must meet clinical procedure success.
Time Frame: Acute: At time of index procedure
Population: Clinical procedure success is computed per subject
Measure: Number; unit: Percentage of success
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2434 | 1216
Percentage of success | 98.6 | 98.1

27. Secondary Outcome: All Myocardial Infarction (MI)
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
Percentage of participants | 1.5 | 2.1

28. Secondary Outcome: All MI
Time Frame: 180 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
Percentage of participants | 1.6 | 2.9

29. Secondary Outcome: All MI
Time Frame: 270 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
Percentage of participants | 1.8 | 3.0

30. Secondary Outcome: All MI
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
Percentage of participants | 1.9 | 3.1

31. Secondary Outcome: All MI
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
Percentage of participants | 2.6 | 3.9

32. Secondary Outcome: All MI
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
Percentage of participants | 3.1 | 4.7

33. Secondary Outcome: All Cause Mortality
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
Percentage of participants | 0.0 | 0.2

34. Secondary Outcome: All Cause Mortality
Time Frame: 180 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
Percentage of participants | 0.5 | 0.6

35. Secondary Outcome: All Cause Mortality
Time Frame: 270 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
Percentage of participants | 0.7 | 0.9

36. Secondary Outcome: All Cause Mortality
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
Percentage of participants | 1.0 | 1.3

37. Secondary Outcome: All Cause Mortality
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
Percentage of participants | 2.1 | 2.7

38. Secondary Outcome: All Cause Mortality
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
Percentage of participants | 3.4 | 5.2

39. Secondary Outcome: Composite Endpoint of All Deaths, All MI, All Revascularizations (DMR)
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
Percentage of participants | 2.4 | 3.6

40. Secondary Outcome: Composite Endpoint of All Deaths, All MI, All Revascularizations (DMR)
Time Frame: 180 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
Percentage of participants | 5.5 | 7.5

41. Primary Outcome: Ischemia Driven Target Lesion Failure (TLF)
Description: Percentage of participants with the determination of TLF. TLF is the composite of cardiac death, target vessel myocardial infarction, and ischemic driven target lesion revascularization (TLR).
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
Percentage of participants | 4.2 | 6.8

42. Secondary Outcome: Composite Endpoint of All Deaths, All MI, All Revascularizations (DMR)
Time Frame: 270 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
Percentage of participants | 7.2 | 9.3

43. Secondary Outcome: Composite Endpoint of All Deaths, All MI, All Revascularizations (DMR)
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
Percentage of participants | 9.0 | 10.5

44. Secondary Outcome: Composite Endpoint of All Deaths, All MI, All Revascularizations (DMR)
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
Percentage of participants | 15.5 | 16.2

45. Secondary Outcome: Composite Endpoint of All Deaths, All MI, All Revascularizations (DMR)
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
Percentage of participants | 21.4 | 22.5

46. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on Academic Research Consortium (ARC) Definition
Description: ARC: Academic Research Consortium-defines ST as a cumulative value at the different time points and with the different seperate time points. Time 0 is defined as the time point after the guiding catheter has been removed. Acute*: 0-24 hours post implantation Subacute*: >24 hours-30 days post Late†: 30 days-1 year post Very late stent thrombosis†: >1 year post
  * Acute/subacute can also be replaced by early ST. Early ST (0-30 days) is currently used in the community.
  † Including "primary" as well as "secondary" late ST; "secondary" late ST is after a target segment revascularization.
Time Frame: 0-30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1221
Percentage of participants | 0.16 | 0.74

47. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on ARC Definition
Description: as for outcome 46
Time Frame: 31-393 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2391 | 1181
Percentage of participants | 0.13 | 0.42

48. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on ARC Definition
Description: as for outcome 46
Time Frame: 0 -393 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2391 | 1181
Percentage of participants | 0.29 | 1.10

49. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on ARC Definition
Description: as for outcome 46
Time Frame: 0-758 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2313 | 1135
Percentage of participants | 0.48 | 1.32

50. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on ARC Definition
Description: as for outcome 46
Time Frame: 0-1123 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2263 | 1098
Percentage of participants | 0.62 | 1.73

51. Secondary Outcome: Protocol Defined Stent Thrombosis Rate
Description: ST will be categorized as acute (≤ 1day), subacute (>1 day to ≤ 30 days) and late (>30 days) and will be defined as any of the following:
  * Clinical presentation of acute coronary syndrome with angiographic evidence of ST
  * In the absence of angiography, any unexplained death, or acute MI (S-T segment elevation or new Q-wave)* in the distribution of the target lesion within 30 days *(Non-specific S-T/T changes, and cardiac enzyme elevations do not suffice) Any thromboses that occur less than 30 days after the index procedure will not be counted as restenosis.
Time Frame: 0-30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1221
Percentage of participants | 0.12 | 0.57

52. Secondary Outcome: Protocol Defined Stent Thrombosis Rate
Description: as for outcome 51
Time Frame: 31-393 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2389 | 1181
Percentage of participants | 0.04 | 0.34

53. Secondary Outcome: Protocol Defined Stent Thrombosis Rate
Description: as for outcome 51
Time Frame: 0-393 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2389 | 1181
Percentage of participants | 0.17 | 0.85

54. Secondary Outcome: Protocol Defined Stent Thrombosis Rate
Description: as for outcome 51
Time Frame: 0-758 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2313 | 1137
Percentage of participants | 0.52 | 1.23

55. Secondary Outcome: Protocol Defined Stent Thrombosis Rate
Description: as for outcome 51
Time Frame: 0-1123 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2266 | 1104
Percentage of participants | 0.79 | 1.99

56. Secondary Outcome: Cardiac Death or Target Vessel MI Rate
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
Percentage of participants | 1.5 | 2.1

57. Secondary Outcome: Cardiac Death or Target Vessel MI Rate
Time Frame: 180 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
Percentage of participants | 1.8 | 2.8

58. Secondary Outcome: Cardiac Death or Target Vessel MI Rate
Time Frame: 270 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
Percentage of participants | 2.1 | 3.0

59. Secondary Outcome: Cardiac Death or Target Vessel MI Rate
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2416 | 1195
Percentage of participants | 2.2 | 3.2

60. Secondary Outcome: Cardiac Death or Target Vessel MI Rate
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
Percentage of participants | 3.2 | 4.3

61. Secondary Outcome: Cardiac Death or Target Vessel MI Rate
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
Percentage of participants | 4.1 | 5.5

62. Secondary Outcome: Ischemia Driven Target Lesion Failure (TLF)
Description: as for outcome 41
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2451 | 1222
Percentage of participants | 1.6 | 2.7

63. Secondary Outcome: Ischemia Driven Target Lesion Failure (TLF)
Description: as for outcome 41
Time Frame: 180 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2435 | 1208
Percentage of participants | 2.5 | 5.1

64. Secondary Outcome: Ischemia Driven Target Lesion Failure (TLF)
Description: as for outcome 41
Time Frame: 270 days
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2419 | 1201
Percentage of participants | 3.4 | 6.1

65. Secondary Outcome: Ischemia Driven Target Lesion Failure (TLF)
Description: as for outcome 41
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2388 | 1190
Percentage of participants | 7.0 | 10.0

66. Secondary Outcome: Ischemia Driven Target Lesion Failure (TLF)
Description: as for outcome 41
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Number analyzed (Participants) | 2348 | 1158
Percentage of participants | 9.5 | 11.9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | XIENCE V® | TAXUS™ EXPRESS 2™
Serious Adverse Events (participants affected / at risk) | 913/2436 | 468/1214
Other Adverse Events (participants affected / at risk) | 762/2436 | 407/1214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE V® (N=2436) | TAXUS™ EXPRESS 2™ (N=1214)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 7 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal symptom (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abscess fungal (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 9 (11) | 5 (5)
Acute prerenal failure (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 11 (12)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 304 (406) | 153 (196)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Aortic aneurysm (Vascular disorders) | 3 (3) | 3 (4)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 6 (6) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arachnoid cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 60 (70) | 43 (48)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial stent insertion (Surgical and medical procedures) | 2 (2) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 1 (1)
Asbestosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (9)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 0 (0)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3)
Blood creatine phosphokinase mb increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2)
Blood glucose flactuation (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 7 (7) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 2 (2) | 1 (1)
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 1 (1)
Cardiac enzymes increased (Investigations) | 4 (4) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 30 (44) | 15 (19)
Cardiac pacemaker insertion (Surgical and medical procedures) | 2 (2) | 0 (0)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 3 (3) | 3 (3)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventriculogram abnormal (Investigations) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Carotid artery disease (Vascular disorders) | 1 (1) | 1 (1)
Carotid artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Vascular disorders) | 9 (9) | 5 (6)
Carotid artery stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 14 (16) | 7 (7)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheter site infection (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 12 (12) | 5 (9)
Central line infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 14 (14) | 12 (12)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Chemotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 8 (8) | 4 (4)
Chest pain (General disorders) | 47 (54) | 24 (29)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 8 (8) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 10 (11)
Clostridial infection (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Computerised tomogram (Investigations) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 3 (3) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery bypass graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 17 (18) | 13 (13)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery perforation (Cardiac disorders) | 4 (4) | 0 (0)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 7 (7) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 3 (4)
Dementia alzheimer's type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Device failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus poor control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic retinal oedema (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ulcer (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 5 (5) | 3 (4)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 6 (6)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1) | 2 (2)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial palsy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 4 (7) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 4 (4) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fibrin d dimer increased (Investigations) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Flank pain (General disorders) | 1 (1) | 0 (0)
Fluid replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture nonunion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 5 (6)
Gangrene (Infections and infestations) | 1 (1) | 1 (3)
Gastric banding (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Vascular disorders) | 47 (57) | 20 (26)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 3 (3)
Gastrooesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gaze palsy (Eye disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Haematemesis (Vascular disorders) | 0 (0) | 1 (1)
Haematochezia (Vascular disorders) | 1 (2) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (7) | 3 (3)
Haemoptysis (Vascular disorders) | 0 (0) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 6 (6) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hemiparesis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 11 (11) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hypoaesthesia facial (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hypotension (Vascular disorders) | 13 (13) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 2 (2) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (2)
Implantable defibrillator insertion (Surgical and medical procedures) | 2 (2) | 1 (1)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infected sebaceous cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (2) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intestinal malrotation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 3 (3) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung lobectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 7 (7)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mechanical complication of implant (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Mediastinoscopy (Investigations) | 1 (1) | 0 (0)
Melaena (Vascular disorders) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 58 (62) | 42 (43)
Myocardial ischemia (Cardiac disorders) | 46 (49) | 18 (20)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 5 (6) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 57 (82) | 28 (30)
Normochromic normocytic anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 (15) | 5 (5)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (5)
Pain (General disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (4) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parathyroid gland operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 8 (10) | 2 (3)
Peripheral vascular disorder (Vascular disorders) | 7 (7) | 1 (1)
Peritoneal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Physiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 4 (5)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 37 (42) | 24 (26)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Vascular disorders) | 3 (3) | 7 (7)
Postoperative abscess (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Vascular disorders) | 0 (0) | 1 (1)
Procedural hypotension (Vascular disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Radiation associated pain (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Rectal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 5 (5) | 2 (2)
Renal artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Renal artery stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal dysplasia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (6) | 5 (5)
Renal failure acute (Renal and urinary disorders) | 20 (23) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal function test abnormal (Investigations) | 1 (1) | 0 (0)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal vessel disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renovascular hypertension (Vascular disorders) | 0 (0) | 1 (1)
Reperfusion injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Vascular disorders) | 6 (6) | 3 (3)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scrotal hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 3 (4) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Subdural hematoma (Vascular disorders) | 2 (3) | 3 (4)
Sudden death (General disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 17 (17) | 7 (8)
Syncope vasovagal (Vascular disorders) | 2 (2) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Transfusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 11 (11) | 7 (7)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (8) | 6 (6)
Urosepsis (Infections and infestations) | 4 (4) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (2) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 21 (21) | 7 (7)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Weight loss poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE V® (N=2436) | TAXUS™ EXPRESS 2™ (N=1214)
Angina pectoris (Cardiac disorders) | 398 (493) | 198 (236)
Back pain (Musculoskeletal and connective tissue disorders) | 193 (194) | 130 (139)
Catheter site haematoma (General disorders) | 177 (181) | 98 (102)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 121 (126) | 64 (67)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will not use Trial related data without written consent of sponsor for any purpose other than Trial completion or generation of publication material. Publication or presentation of results from a trial site are not allowed until publication and/or presentation of multi-center results. Sponsor must receive materials at least 60 days prior to the proposed date of the presentation or the initial submission of proposed publication in order to be reviewed by the sponsor.